CLINICAL TRIAL: NCT00850473
Title: Comparison of Cardiac Positron Emission Tomography/Computed Tomography (PET/CT) With Coronary Angiography (CA) and Intravascular Ultrasound (IVUS) in the Diagnosis and Characterization of Coronary Artery Plaque
Brief Title: PET/CT Study in the Diagnosis of Coronary Plaque
Acronym: PET/CT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sub-investigator left the university
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07-0813; 593F (Other: RDRC); NCT00850473 (Registry Identifier: PET/CT study in the Diagnosis of Coronary Plaque)
Record Dates: First submitted 2009-02-20; First posted 2009-02-25 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Infarction; Coronary Artery Disease; Cardiac Catheterization
Keywords: PET; CT; Heart Attack; Coronary Artery disease; Cardiac Catheterization
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease | interventions — Positron Emission Tomography Computed Tomography; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Positron Emitting Image (Experimental): Patient will have a PET/CT imaging study to determine cardiac stenosis, F-18 FDG and heparin/intralipid infusion and Contrast Dye.will be administered.
  Interventions: Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/CT — Patient will have one imaging modality - a Positron Emitting Tomography CT which includes F-18 FDG and heparin/intralipid infusion and Contrast Dye.
  Other Names: PET/positron Emission Tomography imaging

SUMMARY:
This study is being done to determine if a picture taking test of the heart, positron emission tomography/computed tomography (or cardiac PET/CT), can identify the blockages in the heart arteries that lead to heart attacks when compared to the standard of heart catheterization.

DETAILED DESCRIPTION:
Heart catheterization, in which a thin plastic tube, or catheter, is placed into an artery in the arm or leg and advanced into the heart arteries, is the procedure that you and your doctor have decided to pursue to look for heart artery blockages. It is being performed as part of your standard care and not for research purposes. The research procedure (cardiac PET/CT), which will be performed at a later date is a combination of heart CT (a test that involves the use of x-rays to identify heart artery blockages) and heart PET (an imaging test that uses a radioactive drug to look at how the heart uses fuel (sugar and fats) These tests will be combined (PET/CT) to look for the presence and type of blockage in your heart arteries.

It is important to develop a test that can determine if and what type of blockage you have in your heart arteries as the presence and type of heart artery blockage is a very important predictor of heart attack and death from heart attack.

ELIGIBILITY:
Inclusion Criteria:

* 18 years oof age or older
* referred for cardiac catheterization.
* coronary artery disease that does not need angioplasty.

Exclusion Criteria:

* history of cardiac stents
* bypass surgery
* bad kidney function
* unable to take beta blocker medication
* history of asthma
* allergies to egg containing products
* atrial fibrillation
* pregnancy
* breastfeeding
* overweight by definition of a BMI over 35.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rao, MD, Principal Investigator — Washington University in St. Louis Physicians
Locations (1):
- Cardiovascular Imaging Laboratory, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data available to other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- Positron Emitting Image, F-18 FDG, Contrast Dye: Patient will have a PET/CT imaging study to determine cardiac stenosis, patient will have an injection of F18 FDG to determine the metabolic uptake of the radio-isotope, patient will have contrast dye injected to better visualize the coronary arteries.
Period: Overall Study
Arm/Group | Positron Emitting Image, F-18 FDG, Contrast Dye
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Positron Emitting Image, F18 FDG, Contrast Dye: Patient will have a PET/CT imaging study to determine cardiac stenosis, patient will have an injection of F18 FDG to determine the metabolic uptake of the radio-isotope, patient will have contrast dye injected to better visualize the coronary arteries.
Arm/Group | Positron Emitting Image, F18 FDG, Contrast Dye
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clear Anatomical Landmarks Confirmed by CT
Description: Coronary FDG uptake will be measured at the site of coronary stenosis. The target coronary stenosis will be identified by its proximity to a clear anatomical landmark seen on CT and conventional angiography.
Time Frame: During PET CT scan, an average of 2 hours
Measure: Count of Participants; unit: Participants
Groups:
- Positron Emitting Image: Patient will have a PET/CT imaging study to determine cardiac stenosis
  PET/CT: Patient will have a Positron Emitting Tomography imaging
Arm/Group | Positron Emitting Image
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: During PET CT scan an average of 2 hours
Groups:
- Positron Emitting Image, F18 FDG, Contrast Dye: PET/CT: Patient will have a Positron Emitting Tomography imaging
  Patient will have an injection of F-18-FDG to determine the metabolic uptake of the radioisotope
  Contrast Dye: Patient will be injected with contrast dye to better visualize the coronary arteries
  Heparin/intralipid infusion: Patient will be injected with heparin/intralipid infusion for backgroud myocardial uptake
Arm/Group | Positron Emitting Image, F18 FDG, Contrast Dye
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
There were no limitations or caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes